CLINICAL TRIAL: NCT02578576
Title: The Diagnostic Methods of Crohn's Disease Flare-up Within One Month After Resection
Brief Title: The Diagnostic Methods of Early Postoperative Flare-up of Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, Professor, Jinling Hospital, China
Other Study IDs: DoEPR
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Crohn's Disease
Keywords: Diagnostic Techniques; Digestive System
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients with flare-up: Disease flare-up is demonstrated by coloscopy at one month after resection.
- patients without flare-up: No flare-up is found by coloscopy at one month after resection.

SUMMARY:
Crohn's disease is a chronic inflammatory transmural bowel disorder characterized by high rate of postoperative anastomotic complications and recurrences. Surgery itself can influence immunologic function and trigger inflammatory response, which may result in the flare of Crohn's disease soon after surgery (within one month), especially near the anastomosis. Early flare-up of Crohn's disease can negatively impact the outcomes of operation. However, due to the the complexity of perioperative period and dangerous of invasive examine, it is difficult to distinguish disease flare from postoperative complications.

In this study, the investigators aim to development a diagnostic method of flare-up within one month after surgery, which can help us to detect and then treat disease flare in time.

DETAILED DESCRIPTION:
HBI score, serum CRP, ESR, WBC, Hb, PLT, IL-6，PCT and fecal Calprotectin will be monitored within one month after resection.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing intestinal resection of all macroscopic disease, with an endoscopically accessible anastomosis,

Exclusion Criteria:

* patients have an anastomosis which is endoscopically inaccessible by standard colonoscopy;
* patients withs persisting macroscopic abnormality after surgical resection;
* patients with an end stoma (ileostomy or colostomy);
* patients are not suitable to undergo endoscopy because of co-morbidities or an unwell clinical state;
* patients who are unable to give informed consent;
* patients who are pregnant

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with Crohn's disease
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
flare-up confirmed by coloscopy | one month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute,Jinling Hospital,Nanjing,Jiangsu,China, Nanjing, Jiangsu, China